CLINICAL TRIAL: NCT02391610
Title: A Prospective Population-based Cohort Study That Recruited 16766 Pregnant Women From Six Major Cities of Anhui Province in China
Brief Title: The China-Anhui Birth Cohort Study (C-ABCS)
Status: Completed | Type: Observational
Sponsor: Fangbiao Tao (Other)
Responsible Party: Sponsor-Investigator, Fangbiao Tao, Professor and Dean, Anhui Medical University
Organization: Anhui Medical University (Other)
Other Study IDs: 2008020
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Environmental Exposures; Other Pregnancy With Abortive Outcome; Birth Defects; Children Development
Keywords: birth cohort study; environmental exposures; birth defects; pregnant outcomes; children development
MeSH Terms: conditions — Congenital Abnormalities

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: No intervention

SUMMARY:
The China-Anhui Birth Cohort Study (C-ABCS) was set up to examine the delayed, cumulative and interactive effects of maternal environmental exposures on birth outcomes and children's development. The C-ABCS recruited pregnant women from six major cities of Anhui province, China, between November 2008 and October 2010. A range of data (including demographic, obstetric, occupational, nutritional and psychosocial factors) were collected by both interviews and laboratory tests. In each trimester, women's blood samples were drawn, and pregnancy complications were abstracted from physician's medical records. By the end of 2011, birth outcomes/birth defects were observed/identified by clinicians within 12 months after the delivery of 11 421 singleton live births of six cities and those outcomes among the remaining 2033 live births are still being observed. In addition, 4668 children from Ma'anshan city will be further followed up during the pre-school period till they reach adolescence to obtain the data on familial environmental exposures as well as children's physical, psychological, behavioural and sexual development. The interview data and information on laboratory examinations are available on request from archives in the Anhui Provincial Key Laboratory of Population Health & Aristogenics.

ELIGIBILITY:
Inclusion Criteria:

1. Having been lived in local city at least 6 months;
2. Establishing maternal card in the hospital for the first time;
3. Gestational week ≤ 16 weeks;
4. Willing to have antenatal checkups and childbirth in the hospital where they establish maternal cards.

Exclusion Criteria:

1. Women who have abnormities in speaking and can not complete the survey by themselves;
2. Women with mental disorders;
3. Women who plan to leave local places.

Ages: 17 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The China-Anhui Birth Cohort Study (C-ABCS) is a prospective population-based cohort study that recruited 16766 pregnant women from six major cities of Anhui province in China between November 2008 and October 2010. Six cities were selected for study sites, including Hefei, Ma'anshan, Wuhu, Jieshou, Lu'an and Ningguo. Anhui province is located in the south-east of China. Its socio-economic development is ranked at the mid-level in China. Six cities were selected according to their social and geographic characteristics. These cities are located in Central, Southern and Northern regions of Anhui Province and may represent socio-economic, geographic and cultural variations. In addition, strong local support was one of the important factors to consider in selecting these cities.
Sampling Method: Non-Probability Sample
Enrollment: 16766 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Pregnancy outcomes and birth defects | Up to 12 months of age
  By clinical diagnosis, including abortion/premature birth/prolonged pregnancy/fetal death/stillbirth/live birth, Low birthweight/macrosomia/small for gestation age/large for gestation age, Structural birth defects and functional birth defects

SECONDARY OUTCOMES:
Children's physical development | At ages of 1.5-3 and 4.5-6 years
  Including body height/length, body weight, blood pressure, blood lipoid
Psychological and behavioural development | At ages of 1.5-3 and 4.5-6 years
  cognition, behaviour and temperament
Family environmental exposure | At ages of 1.5-3 and 4.5-6 years
  Eating patterns and parenting style.
Mental health problems | At ages of 1.5-3 & 4.5-6 years
  Mental retardation, attention deficit hyperactivity, disorder, autism spectrum disorders.
Sexual development indicators | At ages of 9-15 years for boys, and 8-14 years for girls
  Secondary sexual characters, Sexual hormones.

REFERENCES:
- [Result] Tao FB, Hao JH, Huang K, Su PY, Cheng DJ, Xing XY, Huang ZH, Zhang JL, Tong SL. Cohort Profile: the China-Anhui Birth Cohort Study. Int J Epidemiol. 2013 Jun;42(3):709-21. doi: 10.1093/ije/dys085. Epub 2012 Jun 21. PMID 22729236